CLINICAL TRIAL: NCT04203173
Title: Financial Incentives And Nurse Coaching to Enhance Diabetes Outcomes - FINANCE-DM
Brief Title: Financial Incentives And Nurse Coaching to Enhance Diabetes Outcomes (FINANCE-DM)-1
Acronym: FINANCE-DM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Leonard Ehianu Egede, Professor & Chair, Department of Medicine, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 1R01DK120861 (NIH)
Record Dates: First submitted 2019-11-26; First posted 2019-12-18 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FINANCE-DM Intervention (Experimental): The FINANCE-DM intervention is comprised of: 1) nurse education, 2) home telemonitoring, and 3) structured financial incentives.
  Interventions: Behavioral: FINANCE-DM
- TIDES Intervention (Active Comparator): Patients randomized to the active comparator group will be assigned the FORA 2-in-1 Telehealth System. A nurse educator will review the glucose and BP readings and use them to tailor and reinforce behavior change.
  Interventions: Behavioral: Active Comparator

INTERVENTIONS:
Behavioral: FINANCE-DM — The FINANCE-DM intervention is comprised of: 1) nurse education, 2) home telemonitoring, and 3) structured financial incentives. Patients randomized to FINANCE-DM will be assigned the FORA 2-in-1 Telehealth System and provided glucose test strips to allow testing at least once a day. BG and BP will be measured daily and results will be uploaded to a secure server. A nurse educator will review the glucose and BP readings and use them to tailor and reinforce behavior change during weekly telephone-delivered diabetes education and skills training session. Participants will also receive financial rewards for: 1) uploading glucose measurements; 2) participating in telephone delivered educational sessions; and 3) absolute percentage drops in HbA1c from baseline at each 3-month follow-up intervals.
  Arms: FINANCE-DM Intervention
Behavioral: Active Comparator — Patients randomized to the active comparator group will be assigned the FORA 2-in-1 Telehealth System and provided glucose test strips to allow testing at least once a day. BG and BP will be measured daily and results will be uploaded to a secure server. A nurse educator will review the glucose and BP readings and use them to tailor and reinforce behavior change during weekly telephone-delivered diabetes education and skills training session.
  Arms: TIDES Intervention

SUMMARY:
The objective of this protocol is to answer the questions: 1) Are financial incentives layered upon nurse education and home telemonitoring superior to nurse education and home telemonitoring alone in improving metabolic control long term? 2) Are the effects of financial incentives on metabolic control sustained once the incentives are withdrawn? and 3) Are financial incentives efficacious within and consistent across racial/ethnic groups? This study provides a unique opportunity to address these gaps in the literature. Investigators propose a randomized controlled trial to test the efficacy of a Financial Incentives And Nurse Coaching to Enhance Diabetes Outcomes (FINANCE-DM) intervention comprised of: 1) nurse education, 2) home telemonitoring, and 3) structured financial incentives; compared to an active control group (nurse education and home telemonitoring alone). The study also will evaluate whether intervention effects are sustained 6 months after the financial incentives are withdrawn (i.e. 18 months post randomization); and whether the intervention is differentially efficacious across racial/ethnic groups.

DETAILED DESCRIPTION:
Study Overview. The overarching aim of this proposal is to test the efficacy of structured financial incentives intervention (FINANCE-DM) comprised of: 1) nurse education, 2) home telemonitoring, and 3) structured financial incentives; compared to an active control group (nurse education and home telemonitoring alone) on glycemic control. The study also will evaluate whether intervention effects are sustained 6 months after the financial incentives are withdrawn (i.e. 18 months post randomization); and whether the intervention is differentially efficacious across racial/ethnic groups. Equal number of patients from three racial/ethnic groups (150 Whites, 150 AAs and 150 HAs, total sample of 450) will be randomized to FINANCE-DM intervention (n=225) or an active comparator group (n=225), so that within each racial/ethnic group, half (75 patients) will be randomized to the FINANCE-DM intervention group and the other half (75 patients) will be randomized to the active comparator group. Primary aims are to test overall efficacy across combined racial/ethnic groups; efficacy within racial/ethnic groups and cost effectiveness for the primary endpoint (glycemic control). Secondary aim is to test efficacy on secondary endpoints including BP, LDL, QOL and self-care behaviors. Each patient will be followed for 12 months (long-term effect) and 18 months (sustainability effect), with study visits at baseline, 3, 6, 9, 12 and 18 months. The FINANCE-DM intervention is comprised of: 1) nurse education, 2) home telemonitoring, and 3) structured financial incentives. The active comparator group will receive the same nurse education and home telemonitoring intervention as the FINANCE-DM group, on the same schedule, and for the same duration . The only difference is that participants will not receive structured financial incentives.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=21 years;
2. Clinical diagnosis of T2DM and HbA1c >=8% at the screening visit;
3. Self-identified as White, AA or HA;
4. Subject must be willing to use the FORA monitoring system for 12 months;
5. Subjects must have access to a landline, Ethernet or cellphone for FORA data uploads for the study period; and 6) Ability to communicate in English.

Exclusion Criteria:

1. Mental confusion on interview suggesting significant dementia;
2. Participation in other diabetes clinical trials;
3. Alcohol or drug abuse/dependency;
4. Active psychosis or acute mental disorder; and
5. Life expectancy <18 months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Glycemic control (HbA1c) | Change from baseline HbA1c at 12 months post intervention follow-ups
  Blood specimens (10cc of blood) will be obtained by trained phlebotomists or nurse for HbA1c.
Resource Utilization and Cost | Change from baseline resource utilization and cost at at 12 months post-intervention follow-ups
  Previously validated questions on resource utilization will be administered. The questionnaires capture information on hospitalizations, physician/professional visits, and medications.

SECONDARY OUTCOMES:
LDL-Cholesterol | Change from baseline cholesterol at at 12 months post intervention follow-ups
  About 10cc of blood will be drawn by trained phlebotomists and sent to the lab for LDL-Cholesterol.
Quality of Life as measured by SF-12 | Change from baseline quality of life measure at at 12 months post intervention follow-ups
  The SF-12 (Ware 1996) is a valid and reliable instrument to measure functional status and reproduces 90% of the variance in PCS-36 and MCS-36 scores.
Systolic and Diastolic Blood Pressure | Change from baseline blood pressure at at 12 months post intervention follow-ups
  Blood pressure readings will be obtained using automated BP monitors (OMRON IntelliSenseTM HEM-907XL). The device will be programmed to take 3 readings at 2-minute intervals, and give an average of the 3 BP readings.
Self-Care Behavior | Change from baseline self-care at at 12 months post intervention follow-ups
  Behavioral skills will be assessed with the Summary of Diabetes Self-Care Activities (SDSCA) scale (Toobert 2000), a brief, validated questionnaire of diabetes self-care. .
Self-Care Behavior Brooks Medication Adherence Scale (BMAS) | Change from baseline self-care at at 12 months post intervention follow-ups
  Medication Adherence will be measured with the 6-item validated self-report Brooks Medication Adherence Scale (BMAS) (Brooks 1994). Each of 6 items measures a specific medication-taking behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard E Egede, MD, MS, Principal Investigator — State University of New York at Buffalo
Locations (1):
- State University of New York at Buffalo, Buffalo, New York, United States

REFERENCES:
- [Background] Egede LE, Walker R, Williams JS, Knapp R, Dismuke CE, Davidson T, Campbell JA. Financial Incentives and Nurse Coaching to Enhance Diabetes Outcomes (FINANCE-DM): a trial protocol. BMJ Open. 2020 Dec 22;10(12):e043760. doi: 10.1136/bmjopen-2020-043760. PMID 33371048
- See also: PDF of study protocol paper — https://bmjopen.bmj.com/content/bmjopen/10/12/e043760.full.pdf